CLINICAL TRIAL: NCT00096421
Title: Tight Glycemic Control in Patients Hospitalized in a Medical-Surgery Intensive Care Unit: A Randomized Study
Brief Title: Tight Glycemic Control in Critical Care Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Pablo Tobón Uribe (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4374-04-13031; 094-2003.
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Critical Illness; Hyperglycemia; Insulin Resistance
Keywords: Critical illness; Critical care; Hyperglycemia; Intensive care; Intensive Care Units; Insulin resistance; Intensive insulin therapy; Conventional insulin therapy
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Insulin Resistance

INTERVENTIONS:
Behavioral: Tight control of blood glucose levels
Behavioral: Conventional control of glucose levels

SUMMARY:
The purpose of this study is to evaluate the impact of tight control of serum glucose levels with an intensive insulin treatment in patients hospitalized in an intensive care unit with medical and surgical patients.

DETAILED DESCRIPTION:
Reduction of morbidity-mortality in critical care patients with tight glycemic control had been proven in surgical patients only.

Study Hypothesis: In critical care patients, medical or surgical, a glucose serum level between 80 - 110 mg/dL means a lower mortality than patients with glucose levels of more than 110 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age or older,
* Probability of staying in critical care for more than 48 hours,
* Agreement with the informed consent.

Exclusion Criteria:

* Pregnancy,
* Participating in other trials,
* Diabetic keto-acidosis or diabetic hyperosmolar state,
* Moribund
* Do-not-resuscitate orders,
* Reentry to the critical care unit of the same patient.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504
Dates: Start 2003-07; Study Completion 2006-09

PRIMARY OUTCOMES:
Mortality in the next 28 days

SECONDARY OUTCOMES:
Mortality during intensive care
Mortality overall in-hospital
Mortality among patients who remained in the intensive care unit for more than five days
Infections incidence in the critical care unit: nosocomial pneumonia, urinary tract infection and catheter related infection
Length of stay in the unit
Days of ventilatory support
Acute renal failure requiring dialysis or hemofiltration
The median number of red-cell transfusions
SOFA score
Critical-illness polyneuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Gisela D De La Rosa, MD, Principal Investigator — Hospital Pablo Tobon Uribe
Locations (1):
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia